CLINICAL TRIAL: NCT04669847
Title: The Effects of Trunk Exercises on Upper Extremity and Respiratory Functions in Duchenne Muscular Dystrophy
Brief Title: The Effects of Trunk Exercises on Upper Extremity and Respiratory Functions in DMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gokce Yagmur Gunes Gencer (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Sponsor-Investigator, Gokce Yagmur Gunes Gencer, Assistant Professor, Akdeniz University
Organization: Akdeniz University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Trunk Training Exercise in DMD
Record Dates: First submitted 2020-01-09; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Muscular Dystrophy, Duchenne; Upper Extremity; Respiratory Functions
Keywords: Duchenne Muscular Dystrophy; Trunk exercise; Trunk control; Upper Extremity; Respiratory functions
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Patients who performed Trunk-oriented exercise program and conventional exercise program
  Interventions: Other: Trunk-oriented exercise program; Other: Conventional exercise program
- Control Group (Experimental): Patients who performed a conventional exercise program
  Interventions: Other: Conventional exercise program

INTERVENTIONS:
Other: Trunk-oriented exercise program — The trunk-oriented exercise program was performed by a physiotherapist two days of the week for 8 weeks.Trunk-oriented exercises were specially adapted to the patient based on the patient's functional status and active participation in the exercises.
  Arms: Study Group
Other: Conventional exercise program — Conventional exercise program was performed daily for 8 weeks, twice a day, on average 45 minutes, each exercise 5-10 repetitions. The program formed stretching exercises, and active or active-assisted strength exercises (upper extremity, lower extremity, abdominal muscles, back muscles).

SUMMARY:
The aim of this study was to investigate the effects of trunk training on trunk control, upper extremity, and pulmonary function in children with Duchenne muscular dystrophy (DMD).

26 children with DMD aged 5-16 were included in the study. They were divided into two groups (study and control). The study group exercised with the trunk-oriented exercise program and the conventional exercise program under the supervision of a physiotherapist, whereas the control group underwent the conventional exercise program under the supervision of their families at home for 8 weeks.

Trunk control, the upper extremity function and respiratory function test were assessed before and after the 8-week exercise program in this study.

DETAILED DESCRIPTION:
This study aimed to investigate the effects of trunk training on trunk control, upper extremity, and pulmonary function in children with Duchenne muscular dystrophy.

26 children with DMD aged 5-16 were included in the study. They were divided into two groups (study and control). The study group (N=13) exercised with the trunk-oriented exercise program and the conventional exercise program under the supervision of a physiotherapist, whereas the control group (N=13) underwent the conventional exercise program under the supervision of their families at home for 8 weeks. The conventional program exercises were taught to patients and their families in the study and control groups. These exercises were performed daily for 8 weeks, twice a day, on average 45 minutes, each exercise 5-10 repetitions. The conventional exercises program formed stretching exercises, and active or active-assisted strength exercises (upper extremity, lower extremity, abdominal muscles, back muscles), and the Trunk-oriented exercises were specially adapted to the patient based on the patient's functional status and active participation in the exercises. Trunk control was assessed using the Trunk Control Measurement Scale, the upper extremity function was assessed using Performance of Upper Limb and respiratory function using the pulmonary function test before and after the 8-week exercise program in this study.

.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Duchenne Muscle Dystrophy
* No injuries and no neurological or orthopedic surgery in the last 6 months
* No other systemic or orthopedic / neurological disorders to prevent exercise

Exclusion Criteria:

-

Ages: 5 Years to 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2018-04-07 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-12-06 (Actual)

PRIMARY OUTCOMES:
Trunk control | 8 weeks
  The trunk control levels of the children were determined according to the Trunk Control Measurement Scale (TCMS). TCMS consists of two sections: static sitting balance and dynamic sitting balance. Dynamic sitting balance is also divided into two subscales: selective movement control and dynamic reaching. The whole scale includes 15 items and all items are scored on a two-, three- or four-point ordinal scale. The total score of the TCMS ranges from 0 to 58, a higher score indicating a better performance of trunk control. TCMS is found to be a reliable and valid assessment to measure trunk control in boys with DMD.
Upper extremity function | 8 weeks.
  Upper Limb Performance was evaluated with The Performance of Upper Limb (PUL) scale. PUL consists of 22 items in total, the items that evaluate upper extremity function at the distal (hand-wrist), middle (elbow), and shoulder levels, and the first item of the scale to evaluate the general upper extremity level. Score options are range from 0-1 to 0-6 depending on the performance of the first item. Each level is evaluated separately, with a maximum score of 16 from the shoulder level, 34 from the middle level, and 24 from the distal level, and a total score of 0-74.
Respiratory function (FEV1) | 8 weeks.
  Respiratory functions were evaluated by pulmonary function tests. Pulmonary function tests were performed in accordance with the American Thoracic Society (ATS) / European Respiratory Society (ERS) criteria, in a sitting position with a computer-compatible spirometer (Cosmed Pony FX machine). Percentages of forced expiratory volume in one second (FEV1) value relative to the expected value was recorded in pulmonary function test.
Respiratory function (FVC) | 8 weeks.
  Respiratory functions were evaluated by pulmonary function tests. Pulmonary function tests were performed in accordance with the American Thoracic Society (ATS) / European Respiratory Society (ERS) criteria, in a sitting position with a computer-compatible spirometer (Cosmed Pony FX machine). Percentages of forced vital capacity (FVC) value relative to the expected value was recorded in pulmonary function test.
Respiratory function (PEF) | 8 weeks.
  Respiratory functions were evaluated by pulmonary function tests. Pulmonary function tests were performed in accordance with the American Thoracic Society (ATS) / European Respiratory Society (ERS) criteria, in a sitting position with a computer-compatible spirometer (Cosmed Pony FX machine). Percentages of peak flow rate (PEF) value relative to the expected value was recorded in pulmonary function test.

CONTACTS AND LOCATIONS:
Overall Officials: GOKCE YAGMUR GUNES GENCER, Principal Investigator — Akdeniz University
Locations (1):
- Gokce Yagmur Gunes Gencer, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No